CLINICAL TRIAL: NCT03824132
Title: IIT2018-05-ASHER-IMPROV2 - LOL: It's All Improv After Cancer!™ - A Randomized Clinical Trial Examining the Impact of an Improvisational Comedy Intervention on Well-Being Among Patients With Cancer
Brief Title: LOL: It's All Improv After Cancer!™
Acronym: IMPROV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arash Asher, MD (Other)
Collaborators: Tower Cancer Research Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Arash Asher, MD, Director, Cancer Rehabilitation & Survivorship, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2018-05-ASHER-IMPROV2
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Psychological Distress
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Improvisational comedy classes
- Waitlist Control Group (Active Comparator)
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Improvisational comedy classes — 6 consecutive improvisational comedy classes
  Arms: Intervention Group
Behavioral: Waitlist control — After 10 week waitlist control, subjects will complete 6 consecutive improvisational comedy classes.
  Arms: Waitlist Control Group

SUMMARY:
This is a 2-arm randomized waitlist controlled trial. A total of 46 of subjects are planned. Subjects will be assigned to the intervention vs. waitlist control group in a randomized fashion. All subjects will complete baseline assessments prior to randomization. Baseline assessments will be completed within two weeks before the start of the improv series. Subjects in the intervention group will complete 6 consecutive improv classes. Patients in the control group will be permitted to complete the improv course (within 10-12 weeks) and follow-up after their 10 week control timeline is complete. Evaluations for the intervention group will be taken at baseline (T0), the last day of class (T1), one month after the last day of class (T2), and 6 months after the last day of class (T3). Evaluations for the waitlist control group will be taken at baseline #1 (T0), 6 weeks after T0 (T1), one month after T1 (T2), first day of class (Baseline 2, T0b), last day of class (T1b), one month after the last day of class (T2b), and 6 months after the last day of class (T3b). Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Total duration of the study is expected to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer stage 1-3 (no distant metastases)
* Completed cancer treatment (including chemotherapy, radiation therapy, biologic treatment, and/or any combination). At time of consent, patient must be at least 2 months (60 days) from their last treatment and no more than 18 months (547 days) post-treatment. Long term hormonal/biologic treatments are ok.
* Adult female age ≥18
* Scores ≤82 on the FACT-G (Patients do not need to maintain score ≤82 after initial screening FACT-G to remain on study)
* Agrees to complete study surveys
* Agrees to attend at least 4 of 6 Improv classes
* English speaking
* Reasonable medical stability (per physician clearance).
* Emotionally stable (per physician clearance) to participate in this series.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Patients who have significant personality disorders or unstable psychiatric disorders that are severe enough to detract from the group process, as determined by their treating physician.
* Patients with severe cognitive impairments, as determined by their treating physician.
* Non-English speakers.
* Patients who have previously participated in an improvisational comedy program in the past year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Overall well-being | 6 weeks
  Change of the Functional Assessment of Cancer Therapy - General (FACT-G) score between the intervention and control groups. Total scores range from 0-108, with higher scores representing better outcomes.

SECONDARY OUTCOMES:
Anxiety | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) Emotional Distress - Anxiety - Short Form 8a score between the intervention and control groups. Total scores range from 8-40, with lower scores representing better outcomes.
Depression | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) Emotional Distress - Depression - Short Form 8a score between the intervention and control groups. Total scores range from 8-40, with lower scores representing better outcomes.
Social Isolation | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) Social Isolation score between the intervention and control groups. Total scores range from 14-70, with lower scores representing better outcomes.
General self-efficacy | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) General Self-Efficacy score between the intervention and control groups. Total scores range from 10-50, with higher scores representing better outcomes.
Self-efficacy for managing emotions | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) Self-Efficacy for Managing Emotions - Short Form 8a score between the intervention and control groups. Total scores range from 8-40, with higher scores representing better outcomes.
Positive psychosocial outcomes of illness | 6 weeks
  Change of the PROMIS (Patient-Reported Outcomes Measurement Information System) Psychosocial Illness Impact - Positive - Short Form 8a score between the intervention and control groups. Total scores range from 32-80, with higher scores representing better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cancer Clinical Trials Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No